CLINICAL TRIAL: NCT04249635
Title: Fetal Programming of Inflammatory Responses and Body Fat by Maternal Obesity: Role of DHA in the Modulation of Epigenetic Markers of Obesity and Metabolic Disease.
Brief Title: Fetal Programming of Immune Response and Body Fat by Maternal Obesity
Acronym: EpiFat
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 1171406
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Body Composition; Obesity
Keywords: Maternal obesity; Body composition; DHA; n-3 LCPUFA
MeSH Terms: conditions — Obesity; Pregnancy in Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood (plasma & serum) Umbilical cord blood (plasma, serum and cord blood mononuclear cells) Placental tissue (biopsies and IHQ) Infant blood samples at 4 months (plasma & serum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Reference Group: Healthy term (> 37 weeks of gestation) newborns of women with pregestational body mass index (BMI) ≥18,5 and <24,9 in the first prenatal visit.
- Maternal obesity (MO) Group: Newborns of women with pregestational BMI ≥30 that received 200 mg/dayDHA supplementation.
  Interventions: Dietary Supplement: DHA
- MO+DHA Group: Newborns from women with pregestational BMI ≥30 that received 800 mg/day DHA supplementation.
  Interventions: Dietary Supplement: DHA

INTERVENTIONS:
Dietary Supplement: DHA — Women received supplementation of Based on Schizochytrium oil, 100% DHA (DSM) from 14 weeks of pregnancy until delivery.
  Groups: MO+DHA Group; Maternal obesity (MO) Group

SUMMARY:
According to the Chilean National Health Survey 2009-2010, 60% of woman in reproductive age are overweight or obese with detrimental consequences on women as well as offspring´s health at long term.

New efforts are required to clarify how increased maternal body fat and obesity previous and during pregnancy impinge an increased cardiometabolic and obesity risk in the progeny. Nowadays it is clear that obesity in adults constitute a chronic state of sub-clinical inflammation characterized by an increased infiltration of monocytes in the adipose tissue as well as an imbalance between increased pro- (M1) and decreased anti- (M2) inflammatory macrophage polarization. Increased inflammatory markers have been found in obese children as young as 3 years of age, but if these markers are present at birth is completely unknown.

Therefore, unveiling the mechanisms implicated in the capability of monocytes to differentiate into pro-inflammatory macrophages at birth would contribute to establish early markers of the potential risk to develop cardio-metabolic diseases. In this context, modulation of M1-M2 polarization seems to be crucial for the development of altered immune response, and this process would be tightly regulated by epigenetic mechanisms.

On the other hand, long chain polyunsaturated fatty acids (LCPUFAs) play a role as precursors of cellular membrane components and modifiers, and as precursors of a plethora of signaling molecules that participates in cardiovascular, metabolic and immune functions. Additionally, DHA regulates gene expression in monocytes and macrophages altering the M1/M2 polarization. The supplementation with DHA in a high risk population of pregestational obese mothers, with known low n-3 intake, would have an important impact on newborn and infant % body fat. An improvement in the n-6/n-3 LCPUFA ratio during pregnancy in humans could represent a primary prevention strategy to revert fetal and neonatal high body fat and a healthy immune system maturation.

The hypothesis of this proposal is that neonates born from obese mothers supplemented with DHA during pregnancy show a reduction in specific markers of high-risk of obesity. These markers would be evidenced as a lower percent of body fat at birth and at 4 months of age, as well as the reversion of functional and epigenetic changes in neonatal monocytes at birth, compared to neonates from obese mothers with low DHA intake.

DETAILED DESCRIPTION:
AIMS:

In neonates born from pregnant women with normal BMI (> 18.5 and <24,9) at the first prenatal visit (<14 weeks of gestation) (Reference Group) and with pre-gestational obesity (BMI >30 Kg/m2) with low (customary) DHA intake (200 mg/day) (MO Group) and pre-gestational obese women supplemented with a high dose of DHA (800 mg/day)(MO+DHA Group) we will:

* Analyze whether maternal DHA supplementation modifies the body composition in neonates and children at 4 months of age.
* Determine whether maternal supplementation with DHA during pregnancy modifies the balance of circulating pro- and anti-inflammatory cytokines and metabolic markers in the mother during pregnancy, the fetus, the placenta and the child at 4 months of age
* Determine whether the response of macrophages to inflammatory mediators associates with altered epigenetic markers in pro- and anti-inflammatory obesity-related-genes in fetal monocytes from obese mothers and if DHA maternal supplementation reverts this phenotype.
* Determine whether maternal obesity translates into changes in the genome-wide DNA methylation profile in fetal monocytes at birth and the impact of maternal DHA supplementation on this epigenetic effect.

METHODOLOGY. The EpiFat study, is a nested cohort in the Maternal obesity control ThrouGh Healthy nuTrition, MIGHT study (PI: Dr. Garmendia NCT02574767). MIGHT study randomized 1000 patients that began their prenatal care before 14 weeks of gestation to one of four parallel study arms: 2 groups received 200 mg/day DHA (based on Schizochytrium oil, 100% DHA, DSM) and 2 groups 800 mg/day DHA, each group had a group with and one without home-based diet and physical activity interventions.

Recruitment and follow up: At admission to the pre-delivery unit, midwives of the Dr. Sótero del Río Hospital invite all the pregnant women who fulfill eligibility criteria to participate in this study and carries out informed consent process.

After recruitment in the EpiFat study, at delivery moment, midwife collect cord blood samples and the placenta tissue. Between 24 to 48 hrs. after delivery, patients are visited by the research midwife to perform anthropometry to the newborn and collect sociodemographic data and clinical information about women health and delivery process.

At 4 months the infants have a visit, in the Research Center in Eating Environment and Prevention of Associated to Nutrition Chronic Diseases (CIAPEC for his Spanish acronym) from the Institute of Nutrition and Food Technology (INTA for his Spanish acronym), to evaluate anthropometry and body composition. In this visit, infant blood samples (5 ml.) and infant health status information are collected. Furthermore, maternal anthropometry is performed, and infant feeding and food frequency surveys are applied to the mother.

Sample Size:

To calculate sample size for body fat percentage (primary outcome) were considered a mean difference of 2.5%, and 3.0 SD that were described by Catalano. Considering a power of 80% and p-value of 0.05, the sample size estimation was 45 subjects per group. The calculation was made using the software Statistics/Data Analysis STATA version 14.0 (Texas, USA). Considering a 20% of loss to follow up the sample size was adjusted to 54 subjects per group.

For the secondary outcome "the epigenetic-driven inflammatory response of neonatal macrophages in vitro" there is no evidence published. However, previous studies from our group have shown that: For % of methylation in the IL-1β promoter, a sample size of 15 newborns per group from normal weight and obese mother was enough to find a statistical difference between the groups, and for IL-10 in macrophages derived from neonatal monocytes 10 subjects per group was needed. Therefore, for these outcomes it was considered a sample size of 15 subjects per group.

NEWBORN AND MATERNAL VARIABLES OF THE STUDY.

The variables included in the study are:

* Variables of newborn/infants: % of body fat & epigenetic-driven inflammatory response in neonatal macrophages.
* Independent variables of the mothers during pregnancy (week 14 and 24-28 of pregnancy): maternal age (years), BMI (kg/m2, classification), weight (kg), height (m), gestational age (week + days), IL-6, IL-1β, TNFα, MCP-1, IL-10 (pg/mL), triglycerides, cholesterol, LDL-cholesterol, VLDL, HDL (all in mg/dl), fasting glycaemia (mg/dL) and insulin (pg/mL), HOMA-IR, adiponectin (ug/mL), plasma levels of DHA (μmol/l).
* Independent variables of the mother at birth: gestational weight gain (kg, classification), type of delivery, hours of labor.
* Independent variables of the newborn: sex, age (weeks at birth, postnatal weeks), weight (g), length (cm), head circumference (cm), ponderal index (kg/m3), weight for gestational age (classification), IL-6, IL-1β, TNFα, MCP-1, IL-10 (pg/mL), plasma levels of DHA (μmol/l), skinfolds (mm) (biceps, triceps, subscapular, suprailiac and tight).
* Other maternal variables: parity, smoking habit, education (years), type of delivery, placental weight (g).

EX VIVO & IN VITRO STUDIES UMBILICAL CORD BLOOD. Umbilical cord blood are collected after delivery and before placental expulsion in Terumo blood collecting bags (40-100 ml) and stored at 4°C until processing (within 1-5 hours after delivery).

DHA LEVELS IN MATERNAL AND FETAL BLOOD: These will be measured in MIGHT Study by gass chromatography.

MONOCYTE ISOLATION, CELL CULTURE AND MACROPHAGE DIFFERENTIATION. Peripheral blood mononuclear cells (PBMC) are separated shortly after birth by Ficoll density gradient using Histopaque-1077 (Sigma-Aldrich, Missouri, US) centrifugation and incubated in RPMI 1640 medium (Sigma-Aldrich, Missouri, US) and seeded at density of 8 to 10 × 106 cells/mL in 100 mm culture dishes at 5% CO2 for 2 h at 37°C. Monocyte identity is assessed by flow cytometry. Monocytes are cultured for 7 days to assess macrophage differentiation. Macrophage polarization is induced by exposing for 24 hours to 100 ng/mL of LPS (SigmaAldrich, Missouri, US) and 20 ng/mL of INFγ (R&D Systems, Minneapolis, US) for M1 or, alternatively, to 20 ng/mL of IL-4 (R&D Systems, Minneapolis, US) for M2 in RPMI medium supplemented with 5% FBS.

Cells are seeded on plastic culture dishes and maintained in a controlled atmosphere incubator, at 37°C with different experimental conditions.

QUANTIFICATION OF PRO- AND ANTI-INFLAMMATORY CYTOKINES, INSULIN, LEPTIN & ADIPONECTIN IN MATERNAL, NEONATAL AND INFANT PLASMA.

These pro and anti-inflammatory mediators, leptin and insulin are quantified using a multiplexed (Bio-Plex platform) immunometric assay (MILLIPLEX xMAP High Sensitivity Human Cytokine Panel, and human metabolic panel, Millipore, Billerica, MA, USA). Quantification of total adiponectin in umbilical cord plasma is done with High Molecular Weight & Total Adiponectin (ALPCO) ELISA kit, according to the manufacturer's instructions.

PREPARATION OF PLACENTAL HOMOGENATES. Placentas are collected at delivery and weighed after trimming of the cord and membranes, immediately placed on ice after delivery and dissected. The chorionic plate, amniotic sac, and decidua removed. Approximately 50 g of villous tissue is cut into small pieces and rinsed with ice-cold physiological saline. Tissue will be placed in ice-cold buffer D [250 mM sucrose, 0.7 μM pepstatin A, 1.6 μM antipain, 80 μM aprotinin, 1 mM EDTA, 10 mM HEPES-Tris (pH 7.4)] at 4°C and homogenized on ice using a polytron. The homogenate is snap-frozen in liquid nitrogen and stored at -80°C until analysis or further processing.

QUANTITATIVE PCR FOR IN VITRO EXPRESSION OF CYTOKINES. RNA is isolated from monocytes using a commercial kit (GenElute, Sigma), according to manufacturer instructions. RT is perform be with the ImProm-II Reverse.

Transcription System (Promega). PCR is carried out using oligonucleotide primers for human TNFα, IL-6, Il-1β, MCP-1 and IL-10. The levels of mRNAs for GADPH, ATP5F1 and RPLP2 are used as internal references. Primers are validated for use: checking amplification, primer concentrations, efficiency primers-HK and stability of HK in experimental conditions. Relative expression of target genes is calculated using the 2-delta delta ct method.

FLOW CYTOMETRY FOR MONOCYTES CHARATERIZATION. The expression of different surface markers is evaluated using flow cytometry, which is performed either in whole blood for identification of monocyte subtypes or in vitro differentiated macrophages for identification of the immunophenotype. Among circulating monocytes (CD86+ cells) classic and non-classic subtypes are assessed according to their surface expression of CD14 and CD16.

Immunophenotype of macrophages (i.e. M1 and M2) are assessed according to the expression of specific markers (e.g. CCR2, CXCL13, CX3CR, CD62L, KLF4, TNFα, NO production). Samples are stained in the laboratory and sent to a Flow Cytometry Facility at Universidad de Chile (CyAnTM ADP analyzer (Beckman Coulter®), within 48 hours.

GLOBAL DNA METHYLOME. The DNA Methylome analysis are done in collaboration with Dr. Graham Burdge and Dr. Karen Lillycrop from Southampton using the Infinium Methylation EPIC BeadChip kit from Illumina.

DNA METHYLATION ANALYSIS. DNA methylation status of the promoter regions (approximately 400 bp from the transcription start site) of the genes coding for TNF-α, IL-6, IL-1β, MCP-1, IL-10, PPARγ and PCG1α will be determined using bisulfite modification coupled to DNA sequencing. Briefly, total DNA extracts from cells will be treated with sodium bisulphite to convert non-methylated cytosine to uracil, and promoter regions will be amplified by PCR using specific according to the strategy used and published by our group. Briefly, one of the PCR primers will be designed including a 5'-biotin tag, which will allow purification the amplicon directly from the PCR mix. Then biotin-containing amplified DNA strand will be transferred to a PyroMark Q96 MD pyrosequencer (Qiagen) for sequencing. Site-specific CpG methylations will be determined as percentage, comparing the signal intensity of non-bisulfite-sensitive CpG (conserved C, methylated CpG) and bisulfite-sensitive CpG (converted C→T, unmethylated CpG).

STATISTICAL ANALYSIS. For descriptive statistics will be applied mean ± SD or median and interquartile range for quantitative variables, and percentage with n for categories. Distributions will be verified with a Shapiro Wilk test. Differences in fat mass and circulating markers will be determined by ANOVA or Kruskal Wallis according to data distribution. Spearman (parametric) or Pearson (no parametric) correlation will be applied to determine the association between dependent and independent (maternal and neonatal) variables. Independent variables will be fitted to logistic and lineal regression models to evaluate interactions as well as to identify confounding factors. For in vitro studies, comparisons between two or more groups will be performed by means of Student's unpaired t-test and analysis of variance (ANOVA), respectively. If the ANOVA demonstrates a significant interaction between variables, post hoc analyses were performed by Dunns when comparing selected groups and multiple-comparison Bonferroni correction test. Data for in vitro responses to cytokines will be fitted to dose-response curves from which maximal response and drug potency (pD2 = -Log EC50) will be obtained. Comparison of curves and maximal responses under different conditions will be analysed by ANOVA. All the analyses will be carried out with the statistical software Graphpad Prism, STATA or SPSS considering a p<0.05 as cut-off for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term (> 37 weeks of gestation) newborns of: women with pregestational BMI ≥18,5 and <24,9 in the first prenatal visit (Reference Group); newborns of women with pregestational BMI ≥30 with customary DHA supplementation (200 mg/day) (Maternal obesity, MO Group); newborns from women with pregestational BMI ≥30 with 800 mg/day DHA supplementation (MO+DHA Group); all with singleton and healthy pregnancies.

Exclusion Criteria:

* Newborns with low birth weight (<2500 g), complications at delivery, or those requiring long-term hospital admission.
* Newborns of women with preexisting diabetes, premature labor, gestational diabetes, preeclampsia, multiple gestation, chronic cardio-respiratory disorder or neurological o genetic defects of the fetus; any high risk pregnancy condition according to national guidelines,

Ages: 24 Hours to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pregnant women of Puente Alto district of Santiago, Chile.
Sampling Method: Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Newborn body fat percentage | 24 hours to 48 hours after birth.
  Percentage of body fat obtained by skinfold measures and calculated using Catalano et al (1996) formula.
Infant body fat | 4 Months of age.
  Percentage and fat mass obtained by Air Displacement Plethysmography (PEA POD)

SECONDARY OUTCOMES:
Epigenetic-driven inflammatory response of neonatal monocytes & macrophages in vitro. | At birth
  Analyze differentially methylated sites in DNA obtained from neonatal monocytes (3 groups)
DHA antiinflammatory effects in neonatal monocytes | At birth
  In vitro antiinflammatory DHA effect on neonatal monocytes

CONTACTS AND LOCATIONS:
Overall Officials: Paola Casanello, Ph.D., Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Red Salud UC Christus Hospital, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided